CLINICAL TRIAL: NCT00285649
Title: Predicting Patients' Response to Spinal Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palmer College of Chiropractic (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U19P3
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Results first posted 2017-07-05 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-07

CONDITIONS: Low Back Pain
Keywords: Spinal Manipulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HVLA-SM (Experimental): HVLA-SM, Experimental, high-velocity low amplitude spinal manipulation
  Interventions: Other: HVLA-SM
- LVVA-SM (Experimental): LVVA-SM, Experimental, low velocity variable amplitude spinal manipulation
  Interventions: Other: LVVA-SM
- Usual Medical Care (Active Comparator): Usual Medical Care, Active Comparator, advice, exercises and medications
  Interventions: Other: Usual Medical Care

INTERVENTIONS:
Other: HVLA-SM — HVLA-SM, Experimental, high-velocity low amplitude spinal manipulation
  Arms: HVLA-SM
Other: LVVA-SM — LVVA-SM, Experimental, low velocity variable amplitude spinal manipulation
  Arms: LVVA-SM
Other: Usual Medical Care — Arm: Active Comparator: Usual Medical Care Usual Medical Care, Active Comparator, advice, exercises and medications (Celebrex, Aleve, Bextra, Naptoxen)
  Arms: Usual Medical Care

SUMMARY:
The purpose of this study is to compare the clinical effectiveness of two types of chiropractic spinal manipulation to conservative medical care for patients at least 55 years old with sub-acute or chronic LBP.

DETAILED DESCRIPTION:
Despite the high prevalence of LBP and the associated economic costs, disability, and lost productivity, and despite the development of several treatment guidelines, one of which recommends chiropractic spinal manipulation for some subgroups of patients with back pain, the management of LBP remains controversial and highly variable across professions and geographic regions. Although one recent publication describes the design of chiropractic and exercise for seniors with low back or neck pain, no published studies, to our knowledge, have assessed the effectiveness of chiropractic manipulation compared to medical care for older adults with sub-acute or chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 55
* Idiopathic mechanical low back pain (LBP) matching classification 1-4 of the Quebec Task Force.
* LBP classified as subacute (onset 4-12 weeks previous) or chronic (onset more than 12 weeks previous), with the current episode occurring at least four weeks prior to the date of contact with the clinic: In order to exclude the greatest proportion of LBP patients that have a favorable natural history of improvement.
* Written Informed Consent
* A minimum baseline score on the Roland Morris Disability Questionnaire (RMQ) of 6 points.

Exclusion Criteria:

* LBP from other somatic tissues as determined by history, examination, and course (e.g. pain referred from visceral conditions).
* LBP diagnosis not meeting Classifications 1 through 4 of the Quebec Task Force, especially the following: low back pain associated with frank radiculopathy defined as typical shooting leg pain; positive straight leg-raising test; an altered lower extremity reflex; a dermatomal sensory deficit; at least one of the following: progressive unilateral muscle weakness or motor loss, or symptoms of cauda equina compression; and CT or MRI evidence of related anatomical pathology (e.g. abnormal disc, stenosis).
* Co-morbid pathology or poor health conditions in patients; Co-morbid conditions and general poor health significantly complicate the prognosis of LBP, and inject a variety of uncontrollable factors in case-management, not to mention experimental analysis and interpretation. Patients who have case histories and physical examination findings indicating other that average good health will be excluded from the study.
* Bone and joint pathology contraindicating patient for SM of the lumbar spine and pelvis: Patients with spinal fractures, tumors, infections, arthropathies, and significant osteoporosis will be referred to appropriate health care.
* Other contraindications for SM of the lumbar spine and pelvis (e.g. bleeding disorders or anticoagulant therapy, extreme obesity).
* Retention of legal advice related to this or a previous LBP episode: Patients with occupational or personal injuries will not be automatically excluded from the study unless they answer yes to a specific question about the retention of legal advice with respect to their LBP episode at the baseline interview.
* Pregnancy: Pregnancy is a contraindication for exposing a patient to ionizing radiation and is a confounding factor in the usual course of LBP.
* Inability to read or verbally comprehend English.
* Clear evidence of narcotic or other drug abuse as determined by history and examination: injects significant confounding factors with respect to internal validity and feasibility.
* Major clinical depression: Patients with scores greater than 17 on the Beck Depression Inventory will be excluded from the study. Patients with evidence of other psychiatric disorders as determined by history and exam will also be excluded.
* Use of manipulative care for any reason within the past 3 months as determined by history: to exclude the possibility of carryover effects.
* Unwillingness to postpone use of all other types of manual treatment for LBP except those provided in the study (including chiropractic and osteopathic SM, physical therapy, and massage) for the duration of the study period: to eliminate confounding effects.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Start 2004-07; Primary Completion 2006-10 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Meeker, DC, M.P.H., Principal Investigator — Palmer Chiropractic College; David Wilder, PhD, Principal Investigator — University of Iowa
Locations (1):
- Palmer Center for Chiropractic Research, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xia T, Long CR, Gudavalli MR, Wilder DG, Vining RD, Rowell RM, Reed WR, DeVocht JW, Goertz CM, Owens EF Jr, Meeker WC. Similar Effects of Thrust and Nonthrust Spinal Manipulation Found in Adults With Subacute and Chronic Low Back Pain: A Controlled Trial With Adaptive Allocation. Spine (Phila Pa 1976). 2016 Jun;41(12):E702-E709. doi: 10.1097/BRS.0000000000001373. PMID 26656041
- [Derived] Hondras MA, Long CR, Haan AG, Spencer LB, Meeker WC. Recruitment and enrollment for the simultaneous conduct of 2 randomized controlled trials for patients with subacute and chronic low back pain at a CAM research center. J Altern Complement Med. 2008 Oct;14(8):983-92. doi: 10.1089/acm.2008.0066. PMID 18990046
- See also: Similar Effects of Thrust and Nonthrust Spinal Manipulation Found in Adults With Subacute and Chronic Low Back Pain: A Controlled Trial With Adaptive Allocation. — https://www.ncbi.nlm.nih.gov/pubmed/26656041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited primarily through direct mail and local media services.
Period: Overall Study
Arm/Group | HVLA-SM | LVVA-SM | Usual Medical Care
Started | 72 | 72 | 48
Completed | 63 | 66 | 42
Not Completed | 9 | 6 | 6
Not completed — Lost to Follow-up | 6 | 4 | 4
Not completed — Withdrawal by Subject | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HVLA-SM | LVVA-SM | Usual Medical Care | Total
Number analyzed (Participants) | 72 | 72 | 48 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (10.0) | 39.3 (8.8) | 40.3 (9.5) | 40.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 22 | 89
  Male | 38 | 39 | 26 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Participant Race: White | 63 | 63 | 43 | 169
  Participant Race: Other | 9 | 9 | 5 | 23
Roland-Morris Disability Questionnaire (RMDQ) [Mean (Standard Deviation); unit: units on a scale] — The RMDQ is a widely used health status measure for low back pain. Scoring of the RMDQ ranges from 0-24, with a higher score indicating an increase in low back pain disability.
  units on a scale | 9.8 (3.6) | 9.5 (3.0) | 9.7 (3.0) | 9.7 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Roland Morris Low Back Pain Disability Questionnaire (RMDQ)
Description: The RMDQ is a widely used health status measure for low back pain. Scoring of the RMDQ ranges from 0-24, with a higher score indicating an increase in low back pain disability. This outcome displays the mean change in RMDQ from baseline to week 3.
Time Frame: Mean change from baseline to week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HVLA-SM | LVVA-SM | Usual Medical Care
Number analyzed (Participants) | 72 | 72 | 48
units on a scale | 4.0 (4.2) | 3.8 (4.1) | 1.0 (3.0)

ADVERSE EVENTS:
Time Frame: From baseline to follow-up at week 3
Description: Any untoward medical occurrence that may present itself during the conduct of the study which may or may not have a causal relationship with the study procedures.
  *The total number of AEs may exceed the total # of people affected because some people experienced multiple AEs.
Groups:
- HVLA-SM*: HVLA-SM, Experimental, high-velocity low amplitude spinal manipulation
  HVLA-SM: HVLA-SM, Experimental, high-velocity low amplitude spinal manipulation
- LVVA-SM*: LVVA-SM, Experimental, low velocity variable amplitude spinal manipulation
  LVVA-SM: LVVA-SM, Experimental, low velocity variable amplitude spinal manipulation
- Usual Medical Care*: Usual Medical Care, Active Comparator, advice, exercises and medications
  Usual Medical Care: Arm: Active Comparator: Usual Medical Care Usual Medical Care, Active Comparator, advice, exercises and medications (Celebrex, Aleve, Bextra, Naptoxen)
Arm/Group | HVLA-SM* | LVVA-SM* | Usual Medical Care*
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72 | 0/48
Other Adverse Events (participants affected / at risk) | 3/72 | 4/72 | 5/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HVLA-SM* (N=72) | LVVA-SM* (N=72) | Usual Medical Care* (N=48)
Low back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 5
Pain/stiffness in the extremities (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No